CLINICAL TRIAL: NCT05354674
Title: Multimodal Deep Learning Signature for Evaluation of Response to Bevacizumab in Patient With Colorectal Cancer Liver Metastasis
Status: Not yet recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xu jianmin, Head of Colorectal Surgery, Fudan University
Other Study IDs: CRC-MULTIMODAL-01 RESEARCH
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer; Liver Metastases
Keywords: colorectal cancer liver metastasis; bevacizumab; radiomics; multimodal
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ARM A: Chemotherapy regimens are determined based on the clinical experience of specialists
  Interventions: Drug: Bevacizumab
- ARM B: Chemotherapy regimens are determined based on the multimodal deep learning signature
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — AEM A：The specialist's decision to add bevacizumab to chemotherapy will be based on their own judgment
  ARM B：The patient's PET/CT imaging, pathology, and clinical information were input into the signature, and the FOLFOX+Bevacizumab regimen was selected when the output label was 1. FOLFOXIRI chemotherapy regimen was selected when the output label was 0

SUMMARY:
Establishment and validation of the deep learning signature of bevacizumab efficacy in initially unresectable CRLM patients

DETAILED DESCRIPTION:
Initially unresectable CRLM patients were included in this study. The tumor response was assessed by local MDT group. The signature will classified patients into responder or non-responder group. We will administer mFOLFOX6+bevacizumab regimen to responders, and FOLFOXIRI regimen to non-responders.

ELIGIBILITY:
Inclusion Criteria:

Age 18-75 years; Histologically proven colorectal adenocarcinoma; Simultaneous liver-limited metastases; Initially unresectable liver metastases determined by a local MDT; Life expectancy of > 3 months; RAS mutation and BRAF V600E wild-type; ECOG 0-1; Available PET/CT imaging before treatment; Available colonoscopy biopsy specimens before treatment

Exclusion Criteria:

Previous systemic treatment for metastatic disease; Previous surgery for metastatic disease; Extrahepatic metastases; Unresectable primary tumor; Major cardiovascular events (myocardial infarction, severe/unstable angina, congestive heart failure, CVA) within 12 months before randomisation; Acute or subacute intestinal obstruction; Second primary malignancy within the past 5 years; Drug or alcohol abuse; No legal capacity or limited legal capacity; Pregnant or lactating women; Uncontrolled hypertension, or unsatisfactory blood pressure control with ≥3 antihypertensive drugs; Peripheral neuropathy;

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Initially unresectable CRLM patients with PET/CT images and colonoscopy biopsy specimens before treatment.
Sampling Method: Non-Probability Sample
Enrollment: 302 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
response rate | 6 months
  response rate will be assessed by local MDT every two months
progression free survival | 3 years
  progression free survival will be assessed by local MDT every two months during

SECONDARY OUTCOMES:
overall survival | 5 years
  overall survival will be assessed by researchers every two months during treatment, and telephone follow-up every three month after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan hospital, Shanghai, Shanghai Municipality, China